CLINICAL TRIAL: NCT00327327
Title: A Phase 1 Trial of Amplimexon® (Imexon, Inj.) Plus Gemcitabine in Advanced, Previously Untreated Pancreatic Adenocarcinoma
Brief Title: Safety Study of Imexon Plus Gemcitabine in Untreated Pancreatic Adenocarcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AmpliMed Corporation (Industry)
Responsible Party: Evan Hersh, VP Medical Affairs, AmpliMed Corporation
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMP-004
Record Dates: First submitted 2006-05-17; First posted 2006-05-18 (Estimated); Last update posted 2010-09-15 (Estimated); Status verified 2010-09

CONDITIONS: Pancreatic Adenocarcinoma
MeSH Terms: interventions — 4-imino-1,3-diazabicyclo(3.1.0)hexan-2-one; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: imexon — 30-60 minutes IV, days 1,8,15 every 28 days
Drug: gemcitabine — 30 minutes IV, days 1,8,15 every 28 days

SUMMARY:
AMP-004 is a Phase 1b dose escalation trial designed to evaluate the safety of the new drug imexon in combination with an approved drug, gemcitabine, for the treatment of patients with previously untreated pancreatic cancer. The treatment consists of dosing with both imexon and gemcitabine on days 1, 8, and 15 of each 28 day cycle. The study is designed to determine the highest doses of the two drugs that can be safely combined together.

ELIGIBILITY:
Inclusion Criteria:

* Inoperable cancer of the pancreas.
* Blood cell counts and blood chemistries in or near normal range.
* Able to perform the activities of daily living.
* A projected life expectancy of at least 2 months.
* If female, neither pregnant nor nursing.
* Willing to use contraceptives to prevent pregnancy.
* No other serious illnesses.
* No other active malignancy.
* No serious infections.
* No current other drug therapy for the cancer or steroid therapy.
* Prior radiation is permitted as is chemotherapy given during radiation or to prevent relapse after surgical removal of the disease.

Exclusion Criteria:

* Prior chemotherapy for metastatic disease.
* Brain metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2004-02; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Determine maximally tolerated dose (MTD) | until MTD reached
determine dose limiting toxicities. | until MTD reached

SECONDARY OUTCOMES:
Changes in plasma thiol levels | until MTD reached
pharmacokinetics | until MTD reached
objective tumor responses. | until MTD reached

CONTACTS AND LOCATIONS:
Overall Officials: Mark Zalupski, MD, Principal Investigator — University of Michigan; Steven Cohen, MD, Principal Investigator — Fox Chase Cancer Center
Locations (9):
- United States (9):
  - Arizona Clinical Research Center, Tucson, Arizona
  - US Oncology Orlando, Cancer Centers of FL, Ocoee, Florida
  - US Oncology Indiana, Indianapolis, Indiana
  - Univ of Michigan, Ann Arbor, Michigan
  - US Oncology Albany, New York Oncology, Albany, New York
  - US Oncology Kettering, Kettering, Ohio
  - Fox Chase Cancer Ctr., Philadelphia, Pennsylvania
  - US Oncology, Virginia Oncology Assoc, Norfolk, Virginia
  - US Oncology Northwest, Northwest Cancer Specialists, Vancouver, Washington

REFERENCES:
- [Result] Cohen SJ, Zalupski MM, Modiano MR, Conkling P, Patt YZ, Davis P, Dorr RT, Boytim ML, Hersh EM. A phase I study of imexon plus gemcitabine as first-line therapy for advanced pancreatic cancer. Cancer Chemother Pharmacol. 2010 Jul;66(2):287-94. doi: 10.1007/s00280-009-1162-y. Epub 2009 Oct 24. PMID 19855966